CLINICAL TRIAL: NCT03538106
Title: Factors Associated With Cesarean Delivery in Women With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0332
Record Dates: First submitted 2017-10-25; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2017-10

CONDITIONS: Pregnant Women; Diabetes Type 1; Cesrean Delivery
Keywords: Cesrean delivery; Risks factors; Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction : Cesarean rate varies from 45% to 73% in the literature in patient with diabetes type 1. Having a prior C-section is the most important risk factor. The aim of this study was to identify risk factor of cesarean in this population.

Methods: This study is an observational, retrospective and single-center study from the hospital of Montpellier. All the pregnancies, planned or not, with subcutaneous insulin infusion or multiple daily injections of insulin, in patients with diabetes type 1 between 2009 and 2015, after 24 weeks of gestation were included. All the data were retrospectively collected by the principal investigator with computer and paper files.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with diabetes type 1
* Pregnancy initiated between 2009 and 2015
* Pregnancy followed up in the universitary hospital center of Montpellier

Exclusion Criteria:

* Women who deliver in an other center
* women with intraperitoneal injections of insulin
* twin gestation
* termination of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnant women with diabetes type 1
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Risk factors associated with a cesarean delivery in patients with diabetes type 1 | 6 years
  he statistical analysis was made with multiple logistic regression using SAS V9.1 and R V3.1.1 programs.

SECONDARY OUTCOMES:
Risk factors associated with a planned cesarean delivery in patients with diabetes type 1 | 6 years
  the statistical analysis was made with multiple logistic regression using SAS V9.1 and R V3.1.1 programs.
Risk factors associated with an emergency cesarean delivery in patients with diabetes type 1 | 6 years
  the statistical analysis was made with multiple logistic regression using SAS V9.1 and R V3.1.1 programs.

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France